CLINICAL TRIAL: NCT05434663
Title: A Phase 4, Open-Label Safety Study of Repeat Doses of SUSTOL in Adult Subjects Receiving Chemotherapy
Brief Title: Safety Study of Repeat Doses of SUSTOL in Adults
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Heron Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HTX-100-403
Record Dates: First submitted 2022-06-22; First posted 2022-06-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Chemotherapy-Induced Nausea and Vomiting (CINV)
Keywords: HTX-100; APF530
MeSH Terms: conditions — Vomiting | interventions — Granisetron; Injections, Subcutaneous

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental)
  Interventions: Drug: SUSTOL

INTERVENTIONS:
Drug: SUSTOL — SUSTOL 10 mg Subcutaneous (SC) on Day 1 of up to 4 cycles.
  Other Names: Granisetron extended-release injection for subcutaneous use

SUMMARY:
This is a repeat-dose, single-arm, open-label study that will evaluate the potential impact of subject-reported injection-site reactions (ISRs) on activities of daily living (ADL) in adult subjects with cancer receiving SUSTOL® (granisetron) extended-release injection, for subcutaneous use for prevention of chemotherapy induced nausea and vomiting (CINV) for up to 4 sequential cycles of chemotherapy (Moderately Emetogenic Chemotherapy [MEC] or Anthracycline and Cyclophosphamide [AC] combination regimen).

ELIGIBILITY:
Inclusion Criteria:

1. Has cancer and is scheduled to receive MEC or AC regimen for at least 4 cycles of chemotherapy, and is prescribed SUSTOL for CINV prevention.
2. Has an Eastern Cooperative Oncology Group performance status of 0 or 1.
3. Has life expectancy of greater than 6 months.
4. Able to receive standardized doses of dexamethasone for the prevention of emesis.
5. Females are eligible only if not pregnant, not lactating, not planning to become pregnant during the study.

Exclusion Criteria:

1. Has hypersensitivity to granisetron, any component of SUSTOL, or any other 5-HT3 Receptor Antagonists.
2. Severe renal impairment (creatinine clearance [CLcr] <30 mL/min).
3. Symptomatic primary or metastatic central nervous system (CNS) disease.
4. Has participated in an interventional clinical study within 30 days of Cycle 1 Day 1.
5. Investigator assessment that subject would not be a good fit for the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-07-06 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with potential impact of subject-reported ISRs on ADL in adult subjects with cancer administered SUSTOL. | 14 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Hattiesburg Clinic Hematology/Oncology, Hattiesburg, Mississippi
  - Gabrail Cancer Center Research, Canton, Ohio